CLINICAL TRIAL: NCT04698460
Title: Functional Efficacy of iFR-guided Hybrid Coronary Revascularization vs Conventional Coronary Artery Bypass Grafting: a Randomized Controlled Study
Brief Title: FUNctional eFficacy of Hybrid coronAry REvascularization
Acronym: FUNFARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The local research project is cancelled because of the organizational issues
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Stanislav Pekarskiy, Lead researcher, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005/e-4
Record Dates: First submitted 2020-12-04; First posted 2021-01-07 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial Revascularization; Coronary Artery Bypass; Internal Mammary-Coronary Artery Anastomosis; Drug-Eluting Stents
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid coronary revascularization (HCR) (Experimental): Patients with multi-vessel CAD randomized to hybrid coronary revascularization
  Interventions: Procedure: Hybrid coronary revascularization
- Conventional coronary artery bypass grafting (CABG) (Active Comparator): Patients with multi-vessel CAD randomized to conventional CABG
  Interventions: Procedure: Coronary artery bypass grafting

INTERVENTIONS:
Procedure: Hybrid coronary revascularization — A staged procedure with a minimally invasive direct coronary artery bypass grafting of left anterior descending artery by left internal mammary artery (LIMA-LAD MIDCAB) at first stage, and percutaneous stenting of iFR-significant lesions in non-LAD arteries at the second stage
  Arms: Hybrid coronary revascularization (HCR)
Procedure: Coronary artery bypass grafting — A conventional procedure of median thoracotomy with on-pump bypass grafting of left anterior descending artery by left internal mammary artery and saphenous vein grafting of circumflex and/or right coronary artery
  Arms: Conventional coronary artery bypass grafting (CABG)

SUMMARY:
The purpose of the study is to compare iFR-guided hybrid coronary revascularization (HCR) and traditional coronary artery bypass grafting (CABG) in terms of a functional efficacy of revascularization assessed by weighted average of iFRs measured 12 month post-procedure in the qualified coronary arteries (all arteries with at least one significant lesion and diameter >1.5 mm at baseline). The true significance of coronary artery disease (CAD) is reflected by the pressure gradients in coronary arteries showing the actual drop in myocardial perfusion whereas the degree of anatomical narrowing in fact only indicates a potential for hemodynamical changes that also depend on vessel compliance, distal vascular resistance, and collateral circulation. Then, the true effect of myocardial revascularization as treatment of CAD should be likewise assessed by measuring residual pressure gradients in coronary arteries remaining after revascularization, i.e. as the functional efficacy in analogy to the functional significance of CAD.

DETAILED DESCRIPTION:
New generation of drug eluting stents (DES) have been shown to have better long-term patency rates than the vein grafts utilized in conventional CABG. Then, it may be expected that hybrid coronary revascularization (HCR) combining minimally invasive direct coronary artery bypass (MIDCAB) grafting of left anterior descending (LAD) artery by left internal mammary artery (LIMA) and stenting of non-LAD coronary arteries with the new generation DESs may have superior efficacy and safety compared to conventional CABG in patients with multivessel coronary artery disease (CAD). The true significance of CAD is reflected by the pressure gradients in coronary arteries that show actual changes in coronary blood flow and myocardial perfusion whereas the degree of anatomical narrowing only indicates a potential for the hemodynamical changes that also depend on vessel compliance, distal vascular resistance, and collateral circulation. Then, the true effect of myocardial revascularization as treatment of CAD should be likewise assessed by measuring residual pressure gradients in coronary arteries after revascularization, i.e. as the functional efficacy in analogy to the functional significance of CAD. For multi-vessel disease the summary hemodynamic effectiveness of revascularization may be captured either by continuous variable, e.g. averaged magnitude of the post-procedural pressure gradients in the qualified arteries or by categorical index, e.g. a relative proportion of the arteries with significant post-procedural pressure gradients among the qualified arteries both preferably weighted for their significance in myocardial blood supply. For comprehensive comparison of the revascularization strategies the qualified arteries should include all arteries/branches that had significant disease at baseline and were amenable to treatment with at least one of the revascularization methods, e.g. with at least one stenosis >70% and diameter >1.5 mm. The categorical measure of the functional efficacy may also be considered a measure of the functional completeness of revascularization in analogy to the conventional anatomical completeness. This functional completeness in terms of removal of all significant pressure gradients in coronary arteries is expected to be superior to anatomical completeness for assessing the procedural success of the intervention because the successful grafting/stent implantation does not guarantee the permanent removal of the pressure gradients, which may still persist due to development of intimal hyperplasia along the suture line of surgical anastomosis or stent underexpansion/edge dissection.

The primary purpose of the study is to assess whether iFR -guided HCR done as the staged procedure with LIMA-LAD MIDCAB at first stage, and percutaneous coronary intervention (PCI) of non-LAD arteries at the second stage, is superior to conventional CABG in terms of the functional efficacy of revascularization assessed by the weighted average of iFRs measured 12 month post-procedure in all coronary arteries with at least one significant stenosis (>70% for CABG group, iFR ≤ 0.89 for iFR-guided HCR) and diameter ≥1.5 mm at baseline. For proximal lesions in major coronary arteries - LAD, circumflex (Cx), and right coronary artery (RCA) - the simple weights 0.5, 0.25, 0.25 will be used, respectively. For other lesions the Duke jeopardy scores will be used instead. Measurement of functional efficacy at 12 month post-procedure will allow assessment of the final result of the intervention after complete vessel healing, endothelialization of the stents, on stable antithrombotic treatment, etc. Also, this study will assess whether achieving the functional completeness of revascularization described above in addition to the anatomical completeness of the procedure may further improve the treatment outcomes in patients with multivessel CAD. Specifically, the investigators will assess the relationship between the functional completeness of the revascularization and the occurrence of the MACCE over 1, 3, and 5 years following randomization in the patients with anatomically complete procedures. Finally, the hypothesis will be tested that iFR-guided HCR has better overall safety than CABG. Whereas, compared to CABG HCR is associated with less frequent perioperative complications, blood transfusions, shorter ICU and hospital stays, these benefits of less invasive treatment may be overridden by the additional complications of stenting, e.g. acute stent thrombosis, dissection, arterial perforation/rupture and others. With iFR guidance of the HCR these additional complications of PCI are expected to be less frequent and the whole procedure - more safe.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Stenosis ≥70% of the LAD and/or ≥50% of left main coronary artery in combination with at least one stenosis ≥70% of the Cx or RCA, suitable for revascularization (decided by a heart team)
* SYNTAX value ≥22.
* Clinical indications for coronary revascularization (angina refractory to optimal medical treatment, ischemia on non-invasive tests, reduced left ventricular ejection fraction)

Exclusion Criteria:

* Previous heart surgery of any kind, including CABG
* Previous surgery involving the left pleural space
* The need for concomitant vascular or other cardiac surgery during index procedure (valve surgery, aortic surgery, left ventricular aneurysmectomy, endarterectomy, etc.)
* Chronic lung disease
* Chronic kidney disease determined as eGFR<60 ml/min/sq.m
* Failure to give informed consent.
* Life expectancy due to non-heart disease is less than 1 year.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Functional efficacy of revascularization | From baseline to 12 month
  Will be assessed as weighted average of the residual (12 month post-procedure) iFRs in coronary arteries that had at least one significant stenosis (>70% for CABG group, iFR ≤ 0.89 for iFR-guided HCR) and diameter ≥1.5 mm at baseline. In case of proximal lesions of LAD, Cx, RCA, the coefficients 0.5; 0.25; 0.25 will be used, respectively. For other lesions Duke jeopardy scores will be used instead (for this scoring, the coronary tree is divided into 6 segments:1) LAD beyond the diagonal branch take-off, 2) major diagonal branch of the LAD, 3) major septal branch of the LAD, 4) Cx beyond the major obtuse margin branch take-off, 5) major obtuse margin branch, and 6) the posterior descending branch of the RCA. Each such segment is assigned 2 points with a possible maximum of 12/12.

SECONDARY OUTCOMES:
Between-group difference in the number of major cardiovascular and cerebral events (MACCE) | From baseline to 12 months, 3, and 5 years
  The components of MACCE will be all-cause mortality, myocardial infarction (MI), stroke, and unplanned coronary revascularization
Between-group difference in the functional efficacy of the revascularization of non-LAD arteries | From baseline to 12 months
  Will be assessed as weighted average of the residual (12 month post-procedure) iFRs in all non-LAD coronary arteries with at least one significant stenosis (>70% for CABG group, iFR ≤ 0.89 for iFR-guided HCR) and diameter ≥1.5 mm at baseline
Between-group difference in the functional completeness of the revascularization | From baseline to 12 months
  The functional completeness will be assessed as the proportion of the coronary arteries with significant iFR at12 month post-procedure among the arteries with at least one significant stenosis (>70% for CABG group, iFR ≤ 0.89 for iFR-guided HCR) and diameter ≥1.5 mm at baseline
Between-group difference in the number of serious adverse events (other than MACCE) | From baseline to 12 months
  Any untoward medical occurrence that is life-threatening, requires inpatient hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability/incapacity
Between-group difference in the frequency of serious adverse events in the peri-operative period | From the day of procedure to one week post-procedure
  Any untoward medical occurrence that is life-threatening, requires prolongation of existing hospitalization, results in persistent or significant disability/incapacity.
  For HCR - a combination of the events during both surgical and endovascular stages (including stent thrombosis, dissections/ perforations/ruptures of coronary arteries, contrast nephropathy, pseudoaneurysms requiring surgical treatment)
Between-group difference in the operation duration | From the time of intubation to the time of discharge from operating room assessed up to 24 hours
  Duration of the operation in minutes
Between-group difference in the mechanical ventilation time | From the intubation to complete withdrawal of ventilation support assessed up to 1 week
  A total inspiratory time when the tidal volume was delivered or the pressure was maintained
Between-group difference in ICU stay | From the time of discharge from operating room to the time of discharge from ICU assessed up to 30 days
  A total time spent in intensive care unit in hours
Between-group difference in the number of patients who undergone re-operation for bleeding | From the index operation to 30 days post-procedure
  Repeat surgery needed for bleeding or cardiac tamponade either before hospital discharge or between hospital discharge and within 30 days of their index operation if discharged earlier than 30 days
Between-group difference in the number of patients who received blood transfusion(s) | From the day of CABG to hospital discharge assessed up to 30 days
  Any transfusion of blood or blood products
Between-group difference in the number of patients with wound infection | From the end of surgery to hospital discharge assessed up to 30 days
  Purulent discharge from the surgical site, wound or drain placed in the wound with at least one of the following signs/symptoms - pain or tenderness, localised swelling, or redness/heat
Between-group difference in hospital stay | From the day of CABG to the discharge after PCI assessed up to 2 months
  A total number of days spent in hospital after surgery including PCI stage
Between-group difference in the number of repeated revascularizations | From baseline to 12 months
  Any surgical or endovascular revascularization
Between-group difference in the number of hospitalizations | From baseline to 12 months follow-up
  Any hospital stay longer than 24 hours
Between-group difference in angina score | 12 months after the procedure
  Canadian Cardiovascular Society Classification
Between-group difference in the quality of life | 12 months after the procedure
  Will be assessed using EQ-5D instrument
Effect of proportion of coronary arteries with significant iFR 12 month post-procedure among the arteries with ≥1 significant stenosis and diameter ≥1.5 mm at baseline on probability of MACCE in patients with anatomically complete procedures | 1, 3, and 5 years following randomization
  Effect of functional completeness of revascularization on occurrence of MACCE evaluated by logistic regression model

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav Pekarskiy, Principal Investigator — Cardiology Research Institute, TNRMC; Yuri Vecherskiy, Principal Investigator — Cardiology Research Institute, TNRMC; Boris Kozlov, Study Director — Cardiology Research Institute, TNRMC
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Centre, Russian Academy of Sciences, Tomsk, Tomsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No